CLINICAL TRIAL: NCT00389363
Title: A Phase II-III Trial Assessing the Efficacy and Safety of Three Doses of the ALK HDM Tablet in House Dust Mite Allergic Patients
Brief Title: Efficacy and Safety Trial of the ALK HDM Tablet in House Dust Mite Allergic Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-02
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: ALK HDM tablet

SUMMARY:
The purpose of the trial is to determine if treatment of asthma patients allergic to house dust mites with the ALK HDM tablet can reduce the need of inhaled corticosteroids (ICS).

ELIGIBILITY:
Inclusion Criteria:

* A history of house dust mite induced asthma
* Use of inhaled corticosteroids (ICS)
* Positive skin prick test to house dust mites
* Positive specific IgE to house dust mites

Exclusion Criteria:

* FEV1 lower than 70%

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Use of inhaled corticosteroid (ICS).

SECONDARY OUTCOMES:
Use of rescue medication and symptoms.
Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Simonsen, MD., Study Director — ALK-Abelló
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Bernstein DI, Kleine-Tebbe J, Nelson HS, Bardelas JA Jr, Sussman GL, Lu S, Rehm D, Svanholm Fogh B, Nolte H. SQ house dust mite sublingual immunotherapy tablet subgroup efficacy and local application site reaction duration. Ann Allergy Asthma Immunol. 2018 Jul;121(1):105-110. doi: 10.1016/j.anai.2018.04.007. Epub 2018 Apr 12. PMID 29656145
- [Derived] Mosbech H, Canonica GW, Backer V, de Blay F, Klimek L, Broge L, Ljorring C. SQ house dust mite sublingually administered immunotherapy tablet (ALK) improves allergic rhinitis in patients with house dust mite allergic asthma and rhinitis symptoms. Ann Allergy Asthma Immunol. 2015 Feb;114(2):134-40. doi: 10.1016/j.anai.2014.11.015. PMID 25624131